CLINICAL TRIAL: NCT00294619
Title: A Phase III, Double-Blind, Randomized, Placebo-Controlled, Parallel-Group, Multicenter Study to Assess Efficacy and Safety of LB03002 Administered Weekly in Adults With Growth Hormone Deficiency.
Brief Title: Treatment of Adults With Growth Hormone Deficiency
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: LG Life Sciences (Industry)
Collaborators: BioPartners GmbH (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BPLG-005
Record Dates: First submitted 2006-02-20; First posted 2006-02-22 (Estimated); Last update posted 2012-10-05 (Estimated); Status verified 2012-10

CONDITIONS: Pituitary Disorders; Adult Growth Hormone Deficiency
Keywords: Growth hormone deficiency
MeSH Terms: conditions — Pituitary Diseases; Dwarfism, Pituitary | interventions — Growth Hormone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- LB03002 (Experimental)
  Interventions: Drug: growth hormone
- Placebo (Placebo Comparator)
  Interventions: Drug: growth hormone

INTERVENTIONS:
Drug: growth hormone — subcutaneous injection, once-weekly

SUMMARY:
The purpose of this study is to evaluate efficacy and safety profile of a new weekly administered growth hormone preparation compared with placebo in adults with growth hormone deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Male or female of at least 23 years and not more than 70 years of age
* GHD of either adult onset(AO)or Childhood onset(CO), either idiopathic or secondary to pituitary disease
* Confirmed diagnosis of GHD defined
* IGF-1 SDS ≤ -1 at screening
* No exposure to rhGH within the last 6 months
* Patients with adequate adrenal function, which is confirmed by ACTH stimulation test at screening; or Patients with known secondary hypoadrenalism on adequate glucocorticoid replacement therapy
* If applicable, hormone replacement therapies for any other hormone deficiencies, adequate and stable for at least 3 months before study entry
* Women of child-bearing potential to be using a reliable method of contraception at the screening and be willing to use it throughout the study
* A negative serum pregnancy test is required at screening for females of child-bearing potential.

Exclusion Criteria:

* History of malignancy other than cranial tumor or leukemia causing GHD or fully treated basal cell carcinoma
* Evidence of active malignancy
* Evidence of growth of pituitary adenoma or other intracranial tumor within the last 12 months, or patients without MRI or CT data to confirm the tumor stability within the last 12 months
* Significant hepatic dysfunction
* Chronic renal impairment
* Clinically significant pulmonary, cardiac, hepatic, renal, or neuromuscular disease
* Prader-Willi syndrome
* Acute severe illness in the last 6 months
* Benign intracranial hypertension
* Active Cushing's syndrome within the last 12 months
* Uncontrolled hypertension
* Patients with overt diabetes mellitus or evidence of persistent impaired glucose tolerance
* Severe psychiatric disease or patients who cannot understand the objective and methods of the study or patients with current alcohol abuse
* Pregnancy or lactation
* Known hypersensitivity to any ingredient of the study drug
* Inability to undergo scanning by dual-energy X ray absorptiometry (DXA) due to a body weight more than 130 kg or in situ internal or external devices known to interfere with DXA scanning
* Weight reducing drugs or appetite suppressants
* Anabolic steroids other than gonadal steroid replacement therapy within 2 months before study entry
* Methylphenidate within 2 months before study entry
* Systemic corticosteroids other than in replacement doses within the 3 months before study entry.
* History of non-compliance with medications, un-cooperativeness or drug abuse
* Patients participating in another study parallel to, or within 6 months prior to study entry, or previous participation in this study
* Patients who are not able to comply with the study protocol for any reason.

Ages: 23 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 147 (Actual)
Dates: Start 2006-04; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

PRIMARY OUTCOMES:
Changes in Fat Mass at the end of 26-week treatment from baseline | 26 weeks

SECONDARY OUTCOMES:
Changes in the following parameters at the end of 26-week treatment from baseline; other body composition parameters, QoL Score, Serum IGF-I, IGFBP-3 levels & SDS, Lipid profile, waist-to-hip ratio | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: HJ Ji, PhD, Study Chair — LG Life Sciences
Locations (1):
- Oregon Health Sciences University, Portland, Oregon, United States